CLINICAL TRIAL: NCT01672671
Title: Identification of BRCA1-associated DNA Repair Dysfunction in Patients With Early Triple Negative Breast Cancer Treated With Neoadjuvant Platinum-based Chemotherapy
Brief Title: BRCA1-associated DNA Repair Dysfunction in Patients With Early Triple Negative Breast Cancer Treated With Neoadjuvant Platinum-based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mona Frolova, Research Associate of Department of Clinical Pharmacology and Chemotherapy, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNNP 001; TNNP 001 (Other: Russian Cancer Research Center named after N.N.Blokhin RAMS)
Record Dates: First submitted 2012-08-16; First posted 2012-08-27 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Early Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Doxorubicin; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant platinum-based chemotherapy (Experimental): Doxorubicin, Paclitaxel, Cisplatin
  Interventions: Drug: Doxorubicin, Paclitaxel, Cisplatin

INTERVENTIONS:
Drug: Doxorubicin, Paclitaxel, Cisplatin — Doxorubicin 25 mg/m2, IV weekly. Number of Cycles: 8 Paclitaxel 100 mg/m2, IV weekly. Number of Cycles: 8. Cisplatin 30 mg/m2, IV weekly. Number of Cycles: 8.

SUMMARY:
The purpose of this study is to assess efficacy of platinum-based neoadjuvant chemotherapy in correlation with BRCA1-associated DNA repair dysfunction in patients with early triple negative breast cancer.

DETAILED DESCRIPTION:
Recent gene expression profiling of breast cancer has identified specific subtypes with clinical, biologic, and therapeutic implications. The basal-like group of tumors is associated with aggressive behavior and poor prognosis, and typically do not express hormone receptors or HER-2 ("triple-negative" phenotype). Therefore, patients with basal-like cancers do not benefit from currently available targeted systemic therapy.

There is a lot of evidence about a link between basal-like breast cancer and BRCA1 deficiency. Many clinical characteristics and molecular features are shared by basal-like breast cancers and tumors that arise in carriers of BRCA1 germline mutations.

Some studies have indicated that BRCA1 mRNA expression was lower in basal-like sporadic cancers than in controls matched for age and grade. BRCA1 is rarely mutated in sporadic breast cancers and, therefore, it is believed that this may be a result of epigenetic mechanisms such as acquired methylation of the BRCA1 gene promoter or a dysfunction in the pathways that regulate BRCA1 expression, such as overexpression of ID4. The profound similarities between hereditary BRCA1-related breast tumors and basal-like tumors strongly implicate a fundamental defect in the BRCA1 or associated DNA-repair pathways (p53, PTEN) in sporadic basal-like tumors.

There is increasing evidence that the BRCA1-related DNA-repair defects, especially defective homologous recombination, determines sensitivity to certain agents, such as platinum salts-based chemotherapy. The complexity in downregulation of BRCA1 expression suggests that these approaches may only be effective in the treatment of a subset of sporadic basal-like cancers. Identification of specific markers for these cancers will be essential to translate an understanding of defective DNA repair into targeted treatments for this poor prognosis subtype.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, age ≥18 years≤75;
2. Histologically confirmed invasive ER-, PR-, and HER2-negative (triple- negative) adenocarcinoma of the breast;
3. Clinical stage T1-2, N0-1, M0.

Exclusion Criteria:

1. Previous treatment for this breast cancer
2. History of malignancy treated with curative intent within the previous 5 years with the exception of skin cancer, cervical carcinoma in situ, or follicular thyroid cancer. Patients with previous invasive cancers (including breast cancer) are eligible if the treatment was completed more than 5 years prior to initiating current study treatment, and there is no evidence of recurrent disease
3. Pregnancy or breast-feeding

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The pathological complete response rate to neoadjuvant platinum-based chemotherapy | after 8 weeks of neoadjuvant chemotherapy
  Pathologic treatment response will be assessed in correlation with BRCA1-associated DNA repair dysfunction signature.

SECONDARY OUTCOMES:
Disease-free survival | 3 years
Clinical responses to neadjuvant chemotherapy | after 8 weeks of neoadjuvant chemotherapy

OTHER OUTCOMES:
Number of patients with 3/4 Grade CTC adverse events to assess toxicity and tolerability of the chemotherapy regimen | after 8 weeks of neadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Russian Cancer Research Center named after N.N.Blokhin RAMS, Moscow, Russia

REFERENCES:
- See also: Breast Cancer, Neoadjuvant Chemotherapy — http://www.ncbi.nlm.nih.gov/pubmed
- See also: Doxorubicin, Paclitaxel, Cisplatin — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp